CLINICAL TRIAL: NCT00134641
Title: A Phase II Study Evaluating Efficacy of the Combination of Gemcitabine and Vinorelbine in Advanced Soft Tissue Sarcoma
Brief Title: Study of Gemcitabine and Vinorelbine in Soft Tissue Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02-282
Record Dates: First submitted 2005-08-24; First posted 2005-08-25 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Sarcoma, Soft Tissue
Keywords: soft tissue sarcoma; metastatic soft tissue sarcoma; gemcitabine; vinorelbine
MeSH Terms: conditions — Sarcoma | interventions — Gemcitabine; Vinorelbine

INTERVENTIONS:
Drug: gemcitabine
Drug: vinorelbine

SUMMARY:
The purpose of this study is to determine if the combination of gemcitabine and vinorelbine is effective in treating patients with advanced soft tissue sarcoma.

DETAILED DESCRIPTION:
Patients will receive both gemcitabine and vinorelbine once a week for two weeks and then one week with no chemotherapy (1 cycle equals 21 days). Gemcitabine and vinorelbine will be administered on day 1 and day 8 of each cycle.

Blood tests will be performed on each day chemotherapy is administered. A CT scan will be done after every 2 cycles (approximately every 6 weeks) to determine the effects of the chemotherapy on the sarcoma.

A physical exam will be performed at the start of chemotherapy and at least every three weeks thereafter.

Patients will remain on this study as long as the disease does not progress or there are no unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of unresectable or metastatic soft tissue sarcoma
* Measurable disease outside of a prior irradiated area
* ECOG performance status 0,1, or 2.
* 0 or 1 prior regimens for advanced disease.
* Adequate end organ function, defined as bilirubin < 1.8; SGOT/SGPT < 2.5 x upper limit of normal (ULN); creatinine < 1.5 x ULN.
* Negative pregnancy test
* Life expectancy of greater than 3 months

Exclusion Criteria:

* Patient has received any investigational agents within 28 days of first day of study drug dosing
* Two or more prior regimens for advanced disease
* Prior gemcitabine or vinorelbine
* Another primary malignancy
* Grade III/IV cardia dysfunction
* Female patients who are pregnant or breast-feeding
* Severe and/or life-threatening medical disease
* Known diagnosis of HIV infection
* Prior chemotherapy within 4 weeks prior to study entry
* Major surgery within 2 weeks prior to study entry
* Known hypersensitivity to either gemcitabine or vinorelbine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-02; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To determine the response of the combination of gemcitabine and vinorelbine in patients with metastatic soft tissue sarcoma

SECONDARY OUTCOMES:
To determine the duration of response and the overall survival of patients with metastatic soft tissue sarcoma being treated with this combination
to evaluate the safety of this combination in this patient population

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne George, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts